CLINICAL TRIAL: NCT00552656
Title: Prospective, Multicenter Study of Firebird Sirolimus-Eluting Stent for Treatment of Complex Coronary Lesions. Clinical and Angiographic Outcomes of FIREMAN Study
Brief Title: Long Term Efficacy and Safety of Firebird Sirolimus-Eluting Stent In Complex Coronary Lesions
Acronym: FIREMAN
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Xijing Hospital (Other)
Collaborators: Air Force Military Medical University, China (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Shanghai MicroPort Medical (Group) Co., Ltd. (Industry); CCheart Consulting Co., Ltd. (Industry)
Responsible Party: Haichang Wang / Director of Department of Cardiology of Xijing Hospital, Xijing Hospital of Fourth Military Military Medical University
Other Study IDs: XJ-20060914
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2008-08

CONDITIONS: Coronary Disease
Keywords: Angioplasty, Transluminal, Percutaneous Coronary; Drug-eluting stents; Treatment Outcome
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: the group of patients with angiographic results of complex coronary lesions(refer to the definition of protocol)are enrolled and given a clinical follow up and angiographic follow up during the following one year.
  Interventions: Device: Firebird(TM) Sirolimus-Eluting Stent

INTERVENTIONS:
Device: Firebird(TM) Sirolimus-Eluting Stent — balloon expandable stent that made of stainless steel.The length is from 13mm-33mm,and the diameter from 2.5mm-4.0mm
  Other Names: sirolimus-eluting stent made in China

SUMMARY:
The purpose of this study is to investigate the long term efficacy and safety of firebird sirolimus-eluting stent for treatment of complex coronary Lesions.

DETAILED DESCRIPTION:
Randomized clinical trials and large-scale registry studies have shown that sirolimus-eluting stents (SESs) decrease major adverse cardiovascular event(MACE)and restenosis rates compared with bare metal stents (BMSs), but relatively small proportion of patients of complex lesions were enrolled in these studies. Moreover,with the increase in complexity of lesions, different DES shows different effects. The long term effects of DES for treatment of complex coronary lesions remains to be established. This study aims to investigate the long term efficacy and safety of Firebird sirolimus-eluting stent implantation in a high-risk population, that is, the patients who had complex coronary lesions, including multivessel diseases,diffuse long lesions, left main lesions, chronic total occlusion, bifurcation lesions, small vessel diseases,severe calcification or angulation lesions, ostial lesions, restenotic lesions after bare metel stent implantation .

ELIGIBILITY:
Inclusion Criteria:

* the patients who have the indication for coronary interventional therapy
* stable angina pectoris (CCS class I II III IV)or unstable angina pectoris (Braunwald class B＆C，I-II) or documented asymptomatic myocardial ischemia
* reference vessel diameter is of 2.5mm to 4.0mm (estimated by investigator)
* significant(>70%) stenosis of target lesion (estimated by investigator)
* angiographic criteria is complex coronary lesions which includes the followings: multivessel lesions(>or=two vessels), diffuse long lesions with length>or=30mm or need two stents overlapped, small vessel lesions(reference vessel diameter<or=2.5mm estimated by investigator), bifurcation lesions need one or two stents and side branch diameter>2.0mm, chronic total occlusion lesions(>3 months), ostial target lesions(including ostial of right coronary artery,left anterior descending artery and left circumflex artery), severe calcification or angulation(location of target lesion at a >45°bend), protected and unprotected left main lesions, restenosis after bare metal stent implantation(core laboratory decision )
* the patients would like to accept the follow-up and sign the informed consent

Exclusion Criteria:

* pregnant or nursing women
* acute myocardial infarction within the preceding one month
* graft lesions after CABG
* implanted other drug-eluting stents at the same time except the designated one
* left ventricle dysfunction with ejection fraction<30%(evaluated by echocardiogram with Simpson's double-chamber method)
* renal dysfunction with serum creatinine level>or=2mg/dl(177umol/L)
* pre-intervention with intravascular brachytherapy or other non-PTCA techniques
* contradictions or allergy to aspirin, heparin, clopidogrel,stainless steel and hypersensitive to contrast media
* anticipated life span < 12 months
* enrollment in other clinical trials at the same time not reaching the primary endpoint and probably interference the present trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the study enrolls a group of high risk population who have angiographic results of complex coronary lesions.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2007-01; Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
cumulative MACE (including cardiac death, non-fatal myocardial infarction and target lesion revascularization) | 3 years

SECONDARY OUTCOMES:
angiographic binary restenosis | 8 months
late loss | 8 months
cumulative target vessel revascularization | 3 years
cumulative in-stent thrombosis | 3 years
cumulative stroke | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Haichang Wang, MD,PhD, Principal Investigator — Director of Department of Cardiology of Xijing Hospital, Fourth Military Medical University
Locations (1):
- Department of Cardiology of Xijing Hospital, Fourth Military Medical University, Xi'an, Shannxi, China

REFERENCES:
- [Background] Lemos PA, Hoye A, Goedhart D, Arampatzis CA, Saia F, van der Giessen WJ, McFadden E, Sianos G, Smits PC, Hofma SH, de Feyter PJ, van Domburg RT, Serruys PW. Clinical, angiographic, and procedural predictors of angiographic restenosis after sirolimus-eluting stent implantation in complex patients: an evaluation from the Rapamycin-Eluting Stent Evaluated At Rotterdam Cardiology Hospital (RESEARCH) study. Circulation. 2004 Mar 23;109(11):1366-70. doi: 10.1161/01.CIR.0000121358.26097.06. Epub 2004 Mar 1. PMID 14993127
- [Derived] Li Y, Li CX, Wang HC, Xu B, Fang WY, Ge JB, Wang WM, Qiao SB, Chen JP, Shen WK, Jiang H, Cong HL, Pu XQ, Qin YW, Jin HG, Cao Y, Huang H. Efficacy and safety of Firebird sirolimus-eluting stent in treatment of complex coronary lesions in Chinese patients: one-year clinical and eight-month angiographic outcomes from the FIREMAN registry. Chin Med J (Engl). 2011 Mar;124(6):817-24. PMID 21518586